CLINICAL TRIAL: NCT00049166
Title: A Phase I Study of OSI-774 in Combination With Standard Fractionation Radiation Therapy in Patients With Oral Cavity or Oropharyngeal Cancer Stage II or III and in Combination With Standard Fractionation Radiation Therapy and Low Dose Daily Cisplatin in Patients With Oral Cavity or Oropharyngeal Cancer Stage III and IV
Brief Title: Erlotinib and Radiation Therapy With or Without Cisplatin in Treating Patients With Mouth or Throat Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03155; NCI-2012-03155 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-5375; JHOC-20020723; JHOC-J0174; 5375 (Other: Johns Hopkins University); 5375 (Other: CTEP); U01CA070095 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Erlotinib Hydrochloride; Cisplatin; Radiotherapy, Intensity-Modulated

ARMS (2):
- Regimen A (erlotinib hydrochloride, IMRT) (Experimental): Patients receive oral erlotinib once daily. Beginning on day 15, patients also undergo IMRT once daily 5 days a week for 7 weeks.
  Patients in both regimens continue to receive erlotinib until the last day of IMRT (patients already in the maintenance phase of this study as of 5/11/04 continue to receive erlotinib once daily for up to 2 years) in the absence of disease progression or unacceptable toxicity.
  In both regimens, cohorts of 3-6 patients receive escalating doses of erlotinib until the MTD is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: erlotinib hydrochloride; Radiation: intensity-modulated radiation therapy; Other: laboratory biomarker analysis
- Regimen B (erlotinib hydrochloride, cisplatin, IMRT) (Experimental): Patients receive oral erlotinib and undergo IMRT as in regimen A. Patients also receive cisplatin IV over 20 minutes on each day of radiotherapy.
  Patients in both regimens continue to receive erlotinib until the last day of IMRT (patients already in the maintenance phase of this study as of 5/11/04 continue to receive erlotinib once daily for up to 2 years) in the absence of disease progression or unacceptable toxicity.
  In both regimens, cohorts of 3-6 patients receive escalating doses of erlotinib until the MTD is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: erlotinib hydrochloride; Drug: cisplatin; Radiation: intensity-modulated radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
  Arms: Regimen B (erlotinib hydrochloride, cisplatin, IMRT)
Radiation: intensity-modulated radiation therapy — Undergo intensity modulated radiation therapy
  Other Names: IMRT
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of combining erlotinib with radiation therapy with or without cisplatin in treating patients who have advanced mouth or throat cancer. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining erlotinib with radiation therapy with or without cisplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determination of the maximally tolerated dose (MTD) of the combination of daily oral OSI-774 and standard fractionation external beam radiation therapy in patients with oral cavity (OC) or oropharyngeal (OP) squamous cell carcinoma (SCC), stage II and III.

II. Determination of the MTD of daily oral OSI-774, low dose daily cisplatin at 6 mg/m^2/day and standard fractionation external beam radiation therapy in patients with oral cavity or oropharyngeal SCC stage III and IV.

III. Determination of the safety of chronic oral dosing of OSI-774 after radiation therapy.

SECONDARY OBJECTIVES:

I. Determination of biological markers of activity of OSI-774 in tumor biopsy specimens from patients with SCC of OC and OP pre and post therapy.

II. Determination of the ability of (18F)-FDG-PET scan to demonstrate biological activity of OSI-774 in previously untreated patients with SCC of the OC and OP and to predict for clinical response.

OUTLINE: This is a multicenter, dose-escalation study of erlotinib. Patients are assigned to 1 of 2 regimens according to disease stage.

Regimen A (patients with stage II [T2, N0] or III [T1-2, N1] disease): Patients receive oral erlotinib once daily. Beginning on day 15, patients also undergo intensity-modulated radiotherapy (IMRT) once daily 5 days a week for 7 weeks.

Regimen B (patients with stage III [T3, N0-1] or IV [T1-4, N2-3, M0 or T4, N0-1, M0] disease): Patients receive oral erlotinib and undergo IMRT as in regimen A. Patients also receive cisplatin IV over 20 minutes on each day of radiotherapy.

Patients in both regimens continue to receive erlotinib until the last day of IMRT (patients already in the maintenance phase of this study as of 5/11/04 continue to receive erlotinib once daily for up to 2 years) in the absence of disease progression or unacceptable toxicity.

In both regimens, cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 30 days and then every 3 months for up to 2 years.

PROJECTED ACCRUAL: A total of 24-48 patients (12-24 per regimen) will be accrued for this study within 6-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical findings consistent with a diagnosis of squamous cell carcinoma of the OC or OP, as determined by the head and neck surgeon, may be recruited to the study prior to diagnostic biopsy; patients must have a histologically confirmed diagnosis of squamous cell carcinoma of OC or OP prior to proceeding with treatment
* Oropharyngeal sites include base of tongue, tonsil, soft palate, and oropharyngeal wall
* Oral cavity sites include oral tongue, buccal mucosa, floor of mouth, retromolar trigone, alveolar ridge, hard palate and mucosal lip
* Patients must be AJCC stage II (T2N0) or III (T1-2N1) (AJCC fifth edition, 1997) for part A of the study, and must be AJCC stage III (T3N 0-1) or IV (T1-4N2-3M0, T4N0-1M0) for part B of the study
* Priority for study entry will be given to patients with easily accessible tumor and who consent to repeat biopsy; study entry will not be restricted to patients who agree to further biopsies; if a patient enrolls on study and later refuses biopsy (excluding diagnostic), he/she may remain on study
* Patients with operable or inoperable tumors will be eligible
* No prior therapy for the tumor, including chemotherapy, radiation therapy, immunotherapy, EGFR targeted therapies, or any other investigational agents
* Prior malignancies of sites other than the head and neck are allowed if disease free interval >= 3 years; basal cell carcinomas of the skin and in situ cervical dysphagias are allowed within this three year interval if completely resected
* Documentation of evaluable tumor less than or equal to four weeks before treatment start
* ECOG performance status = 0, 1 or 2 (Karnofsky >= 60%)
* Life expectancy of greater than or equal to 6 months
* Leukocytes >= 3,000
* Absolute neutrophil count >= 1,500
* Platelets >= 100,000
* Total bilirubin within normal institutional limits unless due to hemolysis or Gilbert's syndrome
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* APTT/INR within normal institutional limits; patients who have abnormalities in APTT/INR that are correctable after administration of vitamin K are eligible
* No uncontrolled diabetes mellitus as glucose must be within a consistently normal range for each patient in order to standardize PET scan interpretations
* No known malabsorption syndrome
* G-tube dependent patients are eligible
* The effects of OSI-774 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with known brain involvement should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to OSI-774 or other agents used in study
* Major surgery or significant traumatic injury occurring within 28 days prior to treatment
* Abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjögren's syndrome), congenital abnormality (e.g., Fuch's dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* Gastrointestinal tract disease resulting in an inability to take oral or enteral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, untreated or new cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because OSI-774 is an epidermal growth factor inhibitor with the potential for teratogenic or abortifacient effects based on the data suggesting that EGFR expression is important for normal organ development; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with OSI-774, breastfeeding should be discontinued if the mother is treated with OSI-774
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with OSI-774; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients on Coumadin are excluded from the study because of reports of interactions between the study drug and Coumadin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-10; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of cisplatin, graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v3.0 | Up to 7 weeks
  Summarized using descriptive statistics.

SECONDARY OUTCOMES:
Time to progression | Up to 2 years
Pharmacokinetics in terms of steady state concentration (Css, min) | Up to 10 weeks
  Relationships between cisplatin and erlotinib hydrochloride steady-state concentrations and toxicity and epidermal growth factor receptor (EGFR) inhibition will be assessed using univariate and multivariate statistical methods.
Percent change in standardized uptake value (SUV) corrected for lean body mass | Up to 14 days
  The pre and post treatment scans will be compared by use of Wilcoxon signed rank test. The relationship between metabolic response and clinical response will be evaluated by use of chi square test or Fisher's exact test as appropriate.
Biological response for each individual patient as defined by determination of the proportional variation of each biomarker | Up to 2 years
  Both pharmacokinetic and pharmacodynamic parameters will be calculated and their relationship fit with flexible regression models.
Relationship between time to treatment failure versus variations in the biomarkers | Up to 2 years
  Analyzed by the Kaplan Meier method or Cox regression models, and tested with a logrank test.
Effect of erlotinib hydrochloride on the EGFR activation and signaling | Up to day 120
  Descriptive statistics (mean +/- standard deviation [SD]) will be used to summarize the data. Differences between pre and post treatment immunohistochemistry (IHC) scored will be compared with a paired-t test.

CONTACTS AND LOCATIONS:
Overall Officials: Maura Gillison, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States